CLINICAL TRIAL: NCT01204515
Title: Abdominal Symptom Phenotype: Pathways to New Biomarkers
Brief Title: Abdominal Symptom Phenotype Study in Children
Acronym: ASPPNB
Status: Completed | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH); University of Washington (Other)
Responsible Party: Principal Investigator, Robert Shulman, M.D., Professor of Pediatrics, Baylor College of Medicine
Other Study IDs: 25755; RC2NR011959 (NIH)
Record Dates: First submitted 2010-09-16; First posted 2010-09-17 (Estimated); Last update posted 2013-02-06 (Estimated); Status verified 2013-02

CONDITIONS: Irritable Bowel Syndrome (IBS)
Keywords: IBS; irritable bowel syndrome; abdominal pain; urgency; bloating; diarrhea; constipation
MeSH Terms: conditions — Irritable Bowel Syndrome; Abdominal Pain; Diarrhea; Constipation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We will be banking DNA for future analysis. The samples will be retained according to the legal and ethical laws.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Girls with IBS: Girls ages 7-12 years who meet Rome III criteria for IBS
- Healthy Girls (controls): Girls ages 7-12 years who are otherwise healthy and have no complaints of stomach pain

SUMMARY:
Children and adults commonly suffer from recurrent abdominal (stomach) pain. One type is called irritable bowel syndrome (IBS). IBS in adults and children is one of the most common and costly health care problems in the US. Some children have pain frequently (recurrent pain) while others rarely have pain. The investigators are conducting this study to help us answer questions about the causes and treatments, and management of IBS in children.

The purpose of this study is to find out if there is more than one type of IBS in children. If there is, this will be important in deciding the best treatments. The investigators also want to learn how children with IBS differ from those who do not have recurrent abdominal (stomach) pain.

DETAILED DESCRIPTION:
Functional gastrointestinal (GI) disorders (FGIDs), in particular irritable bowel syndrome (IBS) in adults and children, are among the most common and costly health care problems in the US. IBS disproportionately affects adult women (10-15% in western nations) and adolescent girls. Yet, health care providers remain challenged to provide effective clinical management. The etiology of IBS is not well defined and likely multi-factorial.

A Need to Define Subgroups of IBS:

This study emerges from the claim that identification of patient subgroups will advance our understanding of IBS and ultimately help develop treatment approaches. Most studies have lumped together patients with IBS into 2 groups (constipation-, diarrhea-predominant) and tested whether they differ from healthy controls. We propose that a paradigm shift is in order. We should recognize that IBS likely has multiple causes and therefore, multiple expressions. We speculate that by understanding better defined patient subgroups and linking them to newer biomarkers or tests, ultimately will further the understanding of the origins and create effective treatments.

ELIGIBILITY:
Inclusion Criteria:

IBS:

* Age 7-12 years
* Females
* Meet criteria for irritable bowel syndrome without evidence of organic disease
* Developmentally normal
* English speaking (as the psychological measures are either not available or validated in Spanish)
* No other chronic, significant (e.g., diabetes, migraines) medical conditions
* No menses

Controls:

* Age 7-12 years
* Females
* No abdominal pain
* No GI or chronic medical conditions (e.g., diabetes)
* Developmentally normal
* English speaking (as the psychological measures are not available or validated in Spanish)
* No menses

Exclusion Criteria:

* Non-english speaking
* Developmentally or cognitively impaired
* Males
* Menses
* No mother in the household for administration of the psychological measures
* Use of any anti-depressants
* History of migraines or chronic pain disorders
* On narcotics for at least 1 week prior to enrollment
* On any NSAIDs or pain reliever for at least 24 hours prior to enrollment
* Sought psychotherapy in past 6 months for abdominal pain

Ages: 7 Years to 12 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Study Population: We are studying only girls in this exploratory study because IBS is more common in girls than boys and the results of these studies can be compared with the results from studies of IBS in adults where the overwhelming number of patients are women.
  Girls who meet the Rome III criteria for IBS or healthy girls with no complaints of stomach pain.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2010-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Compare biomarkers (tests) on girls with and without IBS | Two Days
  Biomarkers: Proteomic analysis of urine samples; Results of video capsule endoscopy (VCE) using the PillCam; Serum lymphocyte activation and cytokine levels (IL-8, IL-10 and IL-12) Responses to DNIC procedure;
Compare the response of stress in girls with and without IBS | One Day
  Salivary cortisol levels prior to and after the diffuse noxious inhibitory control (DNIC) procedure; Psychological characteristics of the child and mother

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Shulman, M.D., Principal Investigator — Baylor College of Medicine - Texas Children's Hospital
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

REFERENCES:
- [Background] Shulman RJ, Eakin MN, Jarrett M, Czyzewski DI, Zeltzer LK. Characteristics of pain and stooling in children with recurrent abdominal pain. J Pediatr Gastroenterol Nutr. 2007 Feb;44(2):203-8. doi: 10.1097/01.mpg.0000243437.39710.c0. PMID 17255832
- [Background] Thakkar K, Gilger MA, Shulman RJ, El Serag HB. EGD in children with abdominal pain: a systematic review. Am J Gastroenterol. 2007 Mar;102(3):654-61. doi: 10.1111/j.1572-0241.2007.01051.x. PMID 17222318
- [Background] Jarrett M, Heitkemper M, Czyzewski DI, Shulman R. Recurrent abdominal pain in children: forerunner to adult irritable bowel syndrome? J Spec Pediatr Nurs. 2003 Jul-Sep;8(3):81-9. doi: 10.1111/j.1088-145x.2003.00081.x. PMID 12942886
- [Background] Burr RL, Motzer SA, Chen W, Cowan MJ, Shulman RJ, Heitkemper MM. Heart rate variability and 24-hour minimum heart rate. Biol Res Nurs. 2006 Apr;7(4):256-67. doi: 10.1177/1099800405285268. PMID 16581896
- [Background] McOmber ME, Shulman RJ. Recurrent abdominal pain and irritable bowel syndrome in children. Curr Opin Pediatr. 2007 Oct;19(5):581-5. doi: 10.1097/MOP.0b013e3282bf6ddc. PMID 17885479
- [Background] Shulman RJ, Eakin MN, Czyzewski DI, Jarrett M, Ou CN. Increased gastrointestinal permeability and gut inflammation in children with functional abdominal pain and irritable bowel syndrome. J Pediatr. 2008 Nov;153(5):646-50. doi: 10.1016/j.jpeds.2008.04.062. Epub 2008 Jun 9. PMID 18538790
- [Background] Lane MM, Weidler EM, Czyzewski DI, Shulman RJ. Pain symptoms and stooling patterns do not drive diagnostic costs for children with functional abdominal pain and irritable bowel syndrome in primary or tertiary care. Pediatrics. 2009 Mar;123(3):758-64. doi: 10.1542/peds.2008-0227. PMID 19254999
- See also: Information about Kids' GI Health — http://www.aboutkidsgi.org/
- See also: Information about Children in Clinical Research Studies — http://www.childrenandclinicalstudies.nhlbi.nih.gov
- See also: Our Research Group's website at Baylor College of Medicine — http://www.bcm.edu/cnrc/kidsabdominalpain